CLINICAL TRIAL: NCT03736382
Title: Mild Intermittent Hypoxia and CPAP: A Multi-pronged Approach to Treat Sleep Apnea in Intact and Spinal Cord Injured Humans
Brief Title: Mild Intermittent Hypoxia and Its Multipronged Effect on Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jason H Mateika, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HL142757, 1 R56HL142757-01; R01HL142757 (NIH); 1R56HL142757-01 (NIH)
Record Dates: First submitted 2018-11-02; First posted 2018-11-09 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea; Spinal Cord Injuries
Keywords: Mild Intermittent Hypoxia; Continuous positive airway pressure therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Spinal Cord Injuries | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group is comprised of participants with OSA and hypertension [either able bodied (Aim 1) or with spinal cord injury (Aim 2)] that will be treated with mild IH and CPAP. In the present proposal, the mild IH protocol will be administered during wakefulness each day for 15 days over a 3-week period to participants that will also be treated with CPAP during sleep. The mild IH protocol will be comprised of a 20-minute baseline period followed by exposure to twelve - two minute episodes of hypoxia [partial pressure of end-tidal oxygen (PETO2) = 50 mmHg]. Each episode will be interspersed with a 2-minute recovery period under normoxic conditions. The PETCO2 will be sustained 2 mmHg above baseline values for the last ten minutes of baseline and throughout the remainder of the protocol.
  Interventions: Other: Mild intermittent hypoxia; Other: Continuous positive airway pressure (CPAP)
- Control Group (Sham Comparator): The control group is comprised of hypertensive OSA participants [either able bodied (Aim 1) or with spinal cord injury (Aim 2)] that will be exposed to a sham protocol in addition to being treated with CPAP during sleep. The sham protocol will be administered during wakefulness for 15 days over a 3-week period. During the sham protocol the participants will be exposed to atmospheric levels of oxygen and carbon dioxide for the duration of the protocol.
  Interventions: Other: Sham protocol; Other: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Other: Mild intermittent hypoxia — Participants will be exposed to twelve two minute episodes of mild intermittent hypoxia 5 days a week for 3 weeks.
  Arms: Experimental Group
Other: Sham protocol — Participants will be exposed to twelve two minute episodes of sham mild intermittent hypoxia (i.e. room air) 5 days a week for 3 weeks.
  Arms: Control Group
Other: Continuous positive airway pressure (CPAP) — All participants will be treated with CPAP each night for a duration of 3 weeks.

SUMMARY:
Mild intermittent hypoxia (IH) initiates sustained increases in chest wall and upper airway muscle activity in humans. This sustained increase is a form of respiratory plasticity known as long-term facilitation (LTF). Repeated daily exposure to mild IH that leads to the initiation of LTF of upper airway muscle activity could lead to increased stability of the upper airway. In line with PI's laboratory's mandate to develop innovative therapies to treat sleep apnea, this increased stability could ultimately reduce the continuous positive airway pressure (CPAP) required to treat obstructive sleep apnea (OSA) and improve compliance with this gold standard treatment. Improved compliance could ultimately serve to mitigate those comorbidities linked to sleep apnea. Moreover, in addition to improving CPAP compliance numerous studies indicate that mild IH has many direct beneficial effects on cardiovascular, neurocognitive and metabolic function. Thus, mild IH could serve as a multipronged therapeutic approach to treat sleep apnea. In accordance with this postulation, our proposal will determine if repeated daily exposure to mild IH serves as an adjunct therapy coupled with CPAP to mitigate associated co-morbidities via its direct effects on a variety of cardiovascular, metabolic and neurocognitive measures and indirectly by improving CPAP compliance. Modifications in autonomic (i.e. sympathetic nervous system activity) and cardiovascular (i.e. blood pressure) function will be the primary outcome measures coupled to secondary measures of metabolic and neurocognitive outcomes.

DETAILED DESCRIPTION:
The dogma over the past 3 decades, particularly in the field of sleep medicine, has been that intermittent hypoxia (IH) is a detrimental stimulus that leads to a number of co-morbidities including autonomic (e.g. increased sympathetic nervous system activity), cardiovascular (e.g. hypertension, atherosclerosis, arterial fibrillation), cognitive (e.g. loss of gray matter, neural injury and impaired neural function coupled to sleepiness) and metabolic dysfunction (dyslipidemia, hyperglycemia, insulin resistance). This belief was based principally on animal studies that employed protocols that were for the most part severe in nature in regards to length and/or intensity of the hypoxic stimulus. However, the elimination of IH in humans with sleep apnea using continuous positive airway pressure (CPAP) has often been ineffective in mitigating the above mentioned co-morbidities. The lack of compliance with CPAP, length of treatment with CPAP (i.e. short durations), and the possibility that IH or other hallmarks of sleep apnea are not the primary mechanism response for the listed co-morbidities, are possible reasons for the absence of improvement in humans.

In contrast to the findings outlined in the previous paragraph, work completed over a similar time frame indicates that some forms of IH may be beneficial in nature. Many studies using a variety of protocols and species, including humans, established that exposure to mild IH initiates sustained increases in the activity of motoneurons, nerves and muscles that contribute to the enhancement of ventilation and the maintenance of upper airway patency. This sustained increase has been termed long-term facilitation (LTF) and this phenomenon has been the focus of PI's research program for two decades. Long-term facilitation is the principle form of respiratory plasticity that we documented in healthy humans, and in humans with obstructive sleep apnea (OSA) and spinal cord injury (SCI). The initiation of this phenomenon is mediated by a number of neuromodulators (e.g. serotonin, adenosine, noradrenaline) that trigger components of at least two cellular pathways, deemed the Q and S pathways, which mediate the phenomenon. Besides the initiation of LTF, studies in rats and humans have provided compelling evidence that mild IH might be cardiovascular (e.g. angiogenesis, reductions in blood pressure, reductions in infarct size), neurocognitive (e.g. brain neurogenesis, reduced oxidative stress and inflammation) and metabolically (e.g. decreased cholesterol, decreased low density and very low lipoprotein, increased high density lipoproteins and reduced hyperglycemia) protective. Many reviews over the past decade, including reviews from PI's laboratory have addressed the underlying physiological cellular mechanisms and the translation to whole animals and humans. Briefly, mild IH may lead to moderate increases in reactive oxygen species. These moderate levels of reactive oxygen species activate transcription factors (e.g. hypoxia-inducible factor 1α, nuclear factor erythroid-derived 2-like 2, GATA binding protein 4) that lead to the induction of many cytoprotective proteins. These proteins serve, for example, to reduce oxidative stress (e.g. superoxide dismutase, glutathione, thioredoxin), inflammation (e.g. inducible nitric oxide synthase), apoptosis (e.g. B-cell lymphoma 2), and promote vasodilation (e.g. heme oxygenase 1) and the formation of blood vessels (e.g. vascular endothelial growth factor). These modifications that ultimately manifest in improved cardiovascular, autonomic and neurocognitive outcomes indicate that beneficial responses can be initiated by IH in a dose dependent fashion without accompanying maladaptive responses. Despite this recognition, the beneficial responses to IH in humans with sleep apnea have not been fully delineated.

Besides these potential beneficial effects it has been established that daily repeated exposure to IH promotes other forms of motor plasticity. Indeed, IH promotes recovery of limb motor function in both rats and humans. Initial studies in humans with SCI revealed that electromyography of the gastrocnemius muscle coupled with measures of ankle torque significantly increased following exposure to brief episodes of IH in humans with SCI. In a subsequent study, exposure to 15 to 90 s episodes of hypoxia each day over 5 consecutive days significantly improved walking speed and duration in 10 meter and 6 minute walking tests in humans with an incomplete SCI. Interestingly, the effect of daily exposure to IH on walking speed was enhanced when combined with 30 minutes of walking each day, which led the authors to conclude that the combined therapies promote greater functional benefits in individuals with incomplete SCI. Thus, daily repeated exposure to IH could have significant therapeutic effects on limb motor function in individuals with SCI accompanied by sleep apnea. Likewise, exposure to this stimulus could promote LTF of upper airway muscle activity leading to reduced therapeutic pressures, improved compliance and enhanced outcome measures as outlined. These possibilities coupled with the direct effects that IH has on those co-morbidities linked to sleep apnea indicates that IH may be effective in mitigating those issues linked to both respiratory and limb motor dysfunction in individuals with sleep apnea and spinal cord injury.

Based on the findings outlined in the previous paragraphs the working hypothesis for the present proposal is that exposure to mild IH leads to LTF of upper airway muscle activity that manifests in increased stability of the upper airway, which could ultimately reduce the CPAP required to treat OSA. As previously reported, a reduction in the therapeutic pressure necessary for the maintenance of airway patency leads to improved comfort and ultimately treatment compliance, which is approximately 40 % amongst users. Indeed, the preliminary data shows that following acute exposure to IH during sleep, and repeated daily exposure to IH during wakefulness, the therapeutic pressure required for the maintenance of upper airway patency was significantly reduced during sleep. The reduced therapeutic pressure was also coupled to a reduction in upper airway resistance and the critical closing pressure. These modifications ultimately led to increased CPAP compliance. The numerous co-morbidities listed in the initial paragraph, which have been linked to hallmarks of sleep apnea (e.g. sleep fragmentation and severe IH), could be significantly improved by increased compliance to CPAP. In addition, as outlined above, IH may directly impact on a variety of co-morbidities associated with sleep apnea independent of CPAP compliance. Collectively, exposure to IH could impact on comorbidities linked to sleep apnea both directly and via improved therapeutic compliance to CPAP.

Aim 1: We will determine if mild IH can serve as an adjunct therapy coupled to CPAP to mitigate associated co-morbidities via its direct effects on a variety of autonomic, cardiovascular, neurocognitive and metabolic measures and indirectly by improving CPAP compliance in able bodied individuals with OSA and hypertension. Our primary outcome variable is blood pressure measured during quiet wakefulness over the 24 hour period. Secondary outcomes include blood pressure measured during sleep over 24 hours, along with the measurement of beat to beat blood pressure, autonomic nervous system activity, blood biomarkers and neurocognitive tests. Additional secondary outcomes include measures of upper airway collapsibility, therapeutic pressure and adherence.

Aim 2: We will employ spinal cord injured participants with OSA and hypertension to determine if mild IH can be coupled with CPAP to mitigate cardiovascular, metabolic and neurocognitive co-morbidities directly, and indirectly by improving CPAP compliance. We will also examine if the mitigation of cardiovascular, metabolic and neurocognitive co-morbidities is accompanied by recovery of respiratory motor function during wakefulness and sleep, and motor limb function during wakefulness following repeated daily exposure to mild IH in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 40 kg/m^2.
* 18 to 60 years old.
* Newly diagnosed sleep apnea (i.e. apnea/hypopnea index < 100 events per hour - average nocturnal oxygen saturation > 85 %) that has not been treated.
* Diagnosed with prehypertension or Stage 1 hypertension as categorized by the American Heart Association
* Not pregnant.
* Normal lung function.
* Minimal alcohol consumption (i.e. no more than the equivalent of a glass of wine/day)
* A typical sleep/wake schedule (i.e. participants will not be night shift workers or have recently travelled across time zones).
* For spinal cord injured participants (Aim-2): incomplete spinal cord lesions at C3 or below and above T12 (greater than 36 mos. post-SCI) without joint contractures but with signs of voluntary ankle, knee and hip movements and the ability to ambulate at least one step without human assistance.

Exclusion Criteria:

* Any disease other than high blood pressure and sleep apnea.
* Medications for high blood pressure and sleep promoting supplements including melatonin
* Current effective CPAP usage (greater than 4 hours per night).
* Night Shift workers or recently traveled across time zones.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure measured during quiet wakefulness over the 24 hour period following mild intermittent hypoxia and sham protocol | Before and after 15 days of exposure to mild intermittent hypoxia or a sham protocol.
  24 hour blood pressure measures will be obtained prior to the beginning and at the end of protocol to quantify blood pressure changes following mild intermittent hypoxia.

SECONDARY OUTCOMES:
Change in blood pressure measured during sleep over 24 hours following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  24 hour blood pressure measures will be obtained prior to the beginning and at the end of protocol to quantify blood pressure changes during sleep following mild intermittent hypoxia.
Change in beat to beat measures of blood pressure following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  Beat to beat blood pressure measures will be obtained to quantify changes induced by MIH+CPAP therapy on beat to beat blood pressure.
Change in sympathetic and parasympathetic nervous system activity following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  Beat to beat blood pressure and electro cardiogram recordings will be obtained to quantify changes in sympathetic and para sympathetic activities due to MIH+CPAP therapy
Change in learning and memory following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  The Buschke Selective Reminding Test will be used to assess changes in learning and memory following mild intermittent hypoxia or sham protocol
Change in attention following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  The Pathfinder Number Test will assess changes in attention following mild intermittent hypoxia or sham protocol
Change in psychomotor function following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  Psychomotor Vigilance Task will be used to measure changes in psychomotor function following mild intermittent hypoxia or sham protocol
Change in daytime sleepiness following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  The Epworth Sleepiness Scale will assess day time sleepiness in mild intermittent hypoxia or sham groups.
Change in overall cognitive function following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  The Mini Mental State Examination will be used to assess five areas of cognition function (i.e. orientation, registration, attention, calculation, recall and language) in mild intermittent hypoxia or sham groups.
Change in respiratory function (for spinal cord injured in Aim-2) | Day 1 and 15 of the protocol
  Measures of respiratory function (respiratory muscle pressure, inspiratory resistive load and magnitude estimation) will be obtained in mild intermittent hypoxia or sham groups.
Change in motor limb function (for spinal cord injured in Aim-2) | Day 1 and 15 of the protocol
  Walking speed using the 10-Meter Walk Test and walking endurance using the 6-Minute Walk Test will be measured in mild intermittent hypoxia or sham groups.
Change in metabolic biomarkers following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  Change in lipid profile and hemoglobin A1C will be used to assess the changes in metabolic biomarkers following mild intermittent hypoxia or sham protocol
Change in inflammatory biomarkers following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  Change in inflammatory biomarkers will be assessed from asymmetric dimethylarginine and high sensitivity C-reactive protein.
Change in angiogenic/vasculogenic biomarkers following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  Change in hypoxia inducible factor 1α and vascular endothelial growth factor will be used to quantify changes in angiogenic/vasculogenic biomarkers.

OTHER OUTCOMES:
Change in upper airway collapsibility following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  Active critical closing pressure will be used to measure changes in upper airway collapsibility
Change in therapeutic pressure following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  Therapeutic pressure for CPAP treatment will be measured at the beginning, mid and end of the protocol.
Change in CPAP treatment adherence following mild intermittent hypoxia and sham protocol | Day 1 and Day 15 of the protocol
  CPAP treatment adherence measured as hours of CPAP use/night will be assessed at the beginning, mid and end of the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jason H Mateika, Ph.D., Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - John D Dingell VA Medical Center, Detroit, Michigan
  - Wayne State University, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No
Publication in peer-reviewed biomedical literature will be the principal means by which final data will be shared. All published papers will be deposited in PubMed Central archive no later than 1 year after publication. When possible, appropriate, and supported by publisher, PI will consider making de-identified data sets available as supplemental material for published manuscripts. Data sets will be uncensored and described in sufficient detail so that others will be able to independently perform statistical analyses to support (or challenge) our conclusions, as well as apply different analytical methods that may give rise to new conclusions and generate new hypotheses. Preservation and access to final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Data will be maintained electronically behind secure Wayne State University firewall. This data will also be kept for six years following the close of study protocol.

REFERENCES:
- [Derived] Panza GS, Puri S, Lin HS, Badr MS, Mateika JH. Daily Exposure to Mild Intermittent Hypoxia Reduces Blood Pressure in Male Patients with Obstructive Sleep Apnea and Hypertension. Am J Respir Crit Care Med. 2022 Apr 15;205(8):949-958. doi: 10.1164/rccm.202108-1808OC. PMID 35015980

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03736382/Prot_SAP_000.pdf